CLINICAL TRIAL: NCT02476214
Title: Comparison of Prenatal Care With Group Guidance to Routine Care for Pregnant Women at Low Risk in Maternal and Child Health Clinics
Brief Title: Comparison of Group Guidance to Routine Care for Pregnant Women at Low Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Arnon D. Cohen, Prof., Meir Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 006/2015ק
Record Dates: First submitted 2015-04-30; First posted 2015-06-19 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Prenatal Care
Keywords: group prenatal care, group guidance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Group prenatal care- receiving prenatal care through a group
  Interventions: Behavioral: group prenatal care
- Control group (No Intervention): Individual prenatal care - receiving regular individual prenatal care

INTERVENTIONS:
Behavioral: group prenatal care — Intervention group Groups of 8-12 women who are in similar week of pregnancy / due date. The first group session will begin at 12-14 week (depends on gestational age at first OBGYN visit). The group meetings will be held once a month until 28 weeks of pregnancy. From 28 weeks and until the end of pregnancy or 40 weeks, it will be held once every two weeks (according to the Ministry of Health guidelines). The last session will be held approximately 6 weeks after birth.
  There will be about 10 group sessions. Each session will be around 90 minutes. At the beginning of every group meeting, the nurse will preform a short anamnesis and measures in private, followed by discussion and guidance. At the end of the session, if needed, women can have private time with the nurse.
  Arms: Intervention group

SUMMARY:
Prenatal care is defined as pregnancy-related health care services provided to a women between conception and delivery. Early, comprehensive prenatal care can promote healthier pregnancies and can reduce the risk of some adverse birth outcomes by detecting and managing preexisting medical conditions, by providing health behavior advice, and by offering a gateway into the health care system for socially disadvantaged women . The customary approach for prenatal care includes routine individual care, which is provided by nurses and physicians in healthcare clinics and hospitals. Since 1995, citizens of Israel, have been entitled to health care services according to the National Health Insurance Law . Israeli citizens are covered by National Health Insurance, and get maternal and child preventive services including prenatal care by local Mother and Child Health Clinics . The prenatal care is individual. A nurse meets with every registered pregnant women, assess the medical and emotional condition and provide guidance related to the pregnancy week of the woman.

Since the 70, a number of group prenatal care intervention programs are described in the literature. Group prenatal care is designed to answer the recommended content for prenatal care for improving the quality of care and resulting in improved pregnancy outcome . The group prenatal care includes three important components: risk assessment. Guidance and support and combines them into the prenatal care22. Creation of the group provides a meeting place for pregnant women. A safe place for sharing and learning from each other and to build a community for mutual support .

The investigators hypothesize that, relative to women who receive standard individual prenatal care, the women who receive group prenatal care will be more likely to:

1. Report higher levels of satisfaction. The investigators also anticipate higher levels of staff satisfaction within the intervention group medical staff.
2. Higher levels of knowledge about pregnancy related issues (e.g., health behaviors during pregnancy, tests during pregnancy).
3. Higher levels of compliance for recommended prenatal care screening tests (e.g., GCT, first and second trimester screening, US)
4. have better perinatal outcomes: better health behaviors during pregnancy (e.g., nutrition, physical activity ext.'), better birth outcomes (e.g., preterm labor, low birthweight,), and better postpartum indicators (e.g., increased breastfeeding);

DETAILED DESCRIPTION:
Prenatal care is defined as pregnancy-related health care services provided to a women between conception and delivery. Early, comprehensive prenatal care can promote healthier pregnancies and can reduce the risk of some adverse birth outcomes by detecting and managing preexisting medical conditions, by providing health behavior advice, and by offering a gateway into the health care system for socially disadvantaged women .

Since 1995, citizens of Israel, have been entitled to health care services according to the National Health Insurance Law . Israeli citizens are covered by National Health Insurance, and get maternal and child preventive services including prenatal care by local Mother and Child Health Clinics . The prenatal care is individual. A nurse meets with every registered pregnant women, assess the medical and emotional condition and provide guidance related to the pregnancy week of the woman. Since the 70', a number of group prenatal care intervention programs are described in the literature. Group prenatal care is designed to answer the recommended content for prenatal care for improving the quality of care and resulting in improved pregnancy outcome . The group prenatal care includes three important components: risk assessment. Guidance and support and combines them into the prenatal care22. Creation of the group provides a meeting place for pregnant women. A safe place for sharing and learning from each other and to build a community for mutual support . In our study, we would like to evaluate feasibility and effectiveness of group Prenatal Care for low risk pregnancies. We hypothesize that, relative to women who receive standard individual prenatal care, the women who receive group prenatal care will be more likely to:

1. Report higher levels of satisfaction. We also anticipate higher levels of staff satisfaction within the intervention group medical staff.
2. Higher levels of knowledge about pregnancy related issues (e.g., health behaviors during pregnancy, tests during pregnancy).
3. Higher levels of compliance for recommended prenatal care screening tests (e.g., GCT, first and second trimester screening, US)
4. have better perinatal outcomes: better health behaviors during pregnancy (e.g., nutrition, physical activity ext.'), better birth outcomes (e.g., preterm labor, low birthweight,), and better postpartum indicators (e.g., increased breastfeeding); The study is an open non-randomized community trial and will include 291 women. 73 of the participants will be in the intervention group. Women who are at high risk pregnancy, under 18 years old or does not speak Hebrew will be excluded. Every women that will arrive to an OBGYN for the first time in the pregnancy, would be asked to join the study. The women who agrees, will be offered either group prenatal care or individual routine prenatal care, depends on their gestational age and the optional group's gestational age. The women can also refuse to be in a group but still be in the control group, if she chooses to. For both arms, data will be collected thru questioners that will be answered at the beginning and at the end of the prenatal care. Data regarding the birth outcomes will be collected from medical files after birth.

In the intervention group: groups of 8-12 women who are in similar week of pregnancy / due date. The first group session will begin at 12-14 week (depends on gestational age at first OBGYN visit). The group meetings will be held once a month until 28 weeks of pregnancy. From 28 weeks and until the end of pregnancy or 40 weeks, it will be held once every two weeks (according to the Ministry of Health guidelines). The last session will be held approximately 6 weeks after birth. There will be about 10 group sessions. Each session will be around 90 minutes. At the beginning of every group meeting, the nurse will preform a short anamnesis and measures in private, followed by discussion and guidance. At the end of the session, if needed, women can have private time with the nurse.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing prenatal care in Maternal and Child Clinics that are a part of the trial
* Age 18+
* Women who speak and understand Hebrew

Exclusion Criteria:

* High risk pregnancies by criteria of Israeli Ministry of Health guidelines

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Care satisfaction | 9 months
  satisfaction form centering care within staff will be assessed by a questionnaire (scale from 1 to 5).
Care satisfaction | 9 months
  satisfaction form centering care within participants, will be assessed by a questionnaire (scale from 1 to 5).
Knowledge | 9 months
  - Levels of knowledge about pregnancy related issues (e.g., health behaviors during pregnancy, tests during pregnancy). will be assessed by a questionnaire (percentage of correct answers).
Adherence to medical recommendations | 9 months
  compliance for recommended prenatal care screening tests
Breastfeeding rates | 9 months
  initiation and duration of breastfeeding (within first 6 weeks after delivery)
Readiness for labor and delivery questionnaire | 9 months
  women's feeling of readiness for delivery

SECONDARY OUTCOMES:
Birth weight | 9 months
  infant weight (in grams) at birth
Birth week | 9 months
  gestational age at birth
Health behaviors during pregnancy | 9 months
  nutrition, physical activity thru the pregnancy, will be assessed by a questionnaire collecting information about behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Clalit Health service, Beersheba, Israel